CLINICAL TRIAL: NCT00259090
Title: A Double-blind, Randomized, Multicentre Trial to Compare the Anti-tumour Effects and Tolerability of a 500 mg Dose of Faslodex (Fulvestrant) Plus Arimidex (Anastrozole) With a 500 mg Dose of Faslodex(Fulvestrant) Alone and With Arimidex(Anastrozole) Alone, in Postmenopausal Women Prior to Surgery for Primary Breast Cancer
Brief Title: Anti-tumour Effects & Tolerability of Faslodex Alone or in Combination With Arimidex in Post Menopausal Women Prior to Surgery for Primary Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6997C00057; 9238IL/0057
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Anastrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Active Comparator): Anastrozole Monotherapy
  Interventions: Drug: Anastrazole
- 2 (Experimental): Fulvestrant Monotherapy
  Interventions: Drug: Fulvestrant
- 3 (Experimental): Anastrozole + Fulvestrant
  Interventions: Drug: Fulvestrant; Drug: Anastrazole

INTERVENTIONS:
Drug: Fulvestrant — 500 mg intramuscular injection
  Other Names: Faslodex; ZD9238
  Arms: 2; 3
Drug: Anastrazole — oral tablet
  Other Names: Arimidex; ZD1033
  Arms: 1; 3

SUMMARY:
To compare the anti-tumour effects as measured by changes in various biomarkers, of a combination of Faslodex and Arimidex with Faslodex alone and Arimidex alone in postmenopausal women patients with primary breast cancer who are awaiting curative-intent surgery.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women.
* Biopsy confirmation of primary breast cancer.
* Oestrogen receptor positive tumour.
* Fit for surgery within one month.
* Written informed consent to participate in the study

Exclusion Criteria:

* Previous treatment with any anti-hormonal therapy for breast cancer.
* Previous radiotherapy to the primary tumour.
* Previous chemotherapy for the primary tumour.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Faslodex Medical Science Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Nottingham, United Kingdom

REFERENCES:
- [Derived] Robertson JF, Dixon JM, Sibbering DM, Jahan A, Ellis IO, Channon E, Hyman-Taylor P, Nicholson RI, Gee JM. A randomized trial to assess the biological activity of short-term (pre-surgical) fulvestrant 500 mg plus anastrozole versus fulvestrant 500 mg alone or anastrozole alone on primary breast cancer. Breast Cancer Res. 2013 Mar 5;15(2):R18. doi: 10.1186/bcr3393. PMID 23497452

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women with oestrogen receptor positive breast cancer, awaiting curative-intent surgery were recruited to 4 medical centres within the UK.
Pre-assignment Details: 121 patients had baseline biopsy and were randomised 1:1:1. 120 patients received 14 to 21 days therapy. Surgery was actually performed between day 13 and 28 and a tumour sample was taken. Safety data is presented for all 120 patients who received therapy. The demography data are summarized for the population who had a usable tumour sample.
Groups:
- Fulvestrant: Fulvestrant 500 mg once monthly injection
- Fulvestrant + Anastrozole: Fulvestrant 500 mg once monthly injection + Anastrozole 1 mg once daily tablet
- Anastrozole: Anastrozole 1 mg once daily tablet
Period: Overall Study
Arm/Group | Fulvestrant | Fulvestrant + Anastrozole | Anastrozole
Started | 35 (Doesn't include protocol deviators, those who didn't complete the study or had missing tumor samples) | 31 (Doesn't include protocol deviators, those who didn't complete the study or had missing tumor samples) | 37 (Doesn't include protocol deviators, those who didn't complete the study or had missing tumor samples)
Completed | 35 | 31 | 37
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant | Fulvestrant + Anastrozole | Anastrozole | Total
Number analyzed (Participants) | 35 | 31 | 37 | 103
Age, Customized [Number; unit: Participants]
  50 - 59 years | 7 (8.5) | 13 (10.5) | 10 (8.7) | 30 (9.0)
  60 - 69 years | 13 | 7 | 14 | 34
  70 - 79 years | 13 | 6 | 9 | 28
  80 - 89 years | 2 | 3 | 2 | 7
  Not available | 0 | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 31 | 37 | 103
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline to Time of Surgery in Oestrogen Receptor (ER) H-score: Antitumour Effects of Fulvestrant, Anastrozole and a Combination of Both as Measured by the ER H-score.
Description: For each sample, the ER H-score is calculated from the percentage of cells staining very weak (+/-); weak (+); moderate (++); or strong (+++) as follows: H-score = [(0.5 x percent +/-) + (1 x percent +) + (2 x percent ++) + (3 x percent +++)]. Range 0-300. The greater the change from baseline (randomization) in ER H-score, the greater the blockage of ER expression and the greater the potential anti-tumour activity. Percentage change from baseline=[(SRG - BL)/BL]x100
Time Frame: Surgery (SRG) was to be performed between days 15 and 22 after baseline (BL)
Measure: Mean (Standard Error); unit: Percentage change from baseline
Arm/Group | Fulvestrant | Fulvestrant + Anastrozole | Anastrozole
Number analyzed (Participants) | 35 | 31 | 37
Percentage change from baseline | -37 (4) | -38 (5) | -7 (6)

2. Primary Outcome: Percentage Change From Baseline to Time of Surgery in Progesterone Receptor (PgR) H-score: Antitumour Effects of Fulvestrant, Anastrozole and a Combination of Both as Measured by the PgR H-score.
Description: For each sample, the PgR H-score is calculated from the percentage of cells staining very weak (+/-); weak (+); moderate (++); or strong (+++) as follows: H-score = [(0.5 x percent+/-) + (1 x percent+) + (2 x percent++) + (3 x percent+++)]. Range 0-300. The greater the change from baseline (randomization in PgR H-score, the greater the blockage of PgR expression and the greater the potential anti-tumour activity. Percentage change from baseline=[(SRG - BL)/BL]x100
Time Frame: Surgery (SRG) was to be performed between days 15 and 22 after baseline (BL)
Population: nine patients with PgR=0 at baseline were excluded from analysis of PgR because the question of medical interest was the effect of treatment on PgR positive patients.
Measure: Mean (Standard Error); unit: Percentage change from baseline
Arm/Group | Fulvestrant | Fulvestrant + Anastrozole | Anastrozole
Number analyzed (Participants) | 33 | 28 | 33
Percentage change from baseline | -31 (8) | -38 (12) | -38 (7)

3. Primary Outcome: Percentage Change From Baseline to Time of Surgery in Ki67 Labelling Index: Antitumour Effects of Fulvestrant, Anastrozole and a Combination of Both as Measured by the Ki67 Labelling Index.
Description: For each sample, the Ki67 labelling index is calculated as the percentage of cells stained positive for Ki67. Range 0-100. The greater the change from baseline (randomization) in Ki67 labelling index, the greater the blockage of Ki67 expression and the greater the potential anti-tumour activity. Percentage change from baseline=[(SRG - BL)/BL]x100
Time Frame: Surgery (SRG) was to be performed between days 15 and 22 after baseline (BL)
Measure: Mean (Standard Error); unit: Percentage change from baseline
Arm/Group | Fulvestrant | Fulvestrant + Anastrozole | Anastrozole
Number analyzed (Participants) | 35 | 31 | 37
Percentage change from baseline | -62 (4) | -68 (6) | -75 (4)

ADVERSE EVENTS:
Arm/Group | Fulvestrant | Fulvestrant + Anastrozole | Anastrozole
Serious Adverse Events (participants affected / at risk) | 0/40 | 3/40 | 2/40
Other Adverse Events (participants affected / at risk) | 18/40 | 13/40 | 17/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant (N=40) | Fulvestrant + Anastrozole (N=40) | Anastrozole (N=40)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0
Unevaluable Event (General disorders) | 0 | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 0 | 1
Procedural Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant (N=40) | Fulvestrant + Anastrozole (N=40) | Anastrozole (N=40)
Constipation (Gastrointestinal disorders) | 3 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3 | 2
Injection Site Rash (General disorders) | 3 | 0 | 0
Unevaluable Event (General disorders) | 3 | 0 | 3
Injection Site Pain (General disorders) | 2 | 1 | 3
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2
Headache (Nervous system disorders) | 3 | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Hot Flush (Vascular disorders) | 7 | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AZ shall have a period of 30 days from receipt of the proposed final manuscript for any publication or other disclosure to review it and may within such time request that submission for publication or disclosure of the manuscript be delayed for no more than an additional 45 days in order for AZ to file patent applications.